CLINICAL TRIAL: NCT03289026
Title: A Multicenter, Open-label Study to Evaluate the Effectiveness and Safety of Aripiprazole in Patients With Acute Episode of Schizophrenia
Brief Title: Pharmacologic Treatment of Acute Episode of Schizophrenia: a Real World Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Si Tianmei, Director of Clinical Psychopharmacology Division, Peking University Sixth Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 320-57-1706-1101-0001
Record Dates: First submitted 2017-09-17; First posted 2017-09-20 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Acute Schizophrenia Episode
Keywords: Aripiprazole; Acute schizophrenia episode; positive symptoms
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- aripiprazole group (Experimental): Patients receive aripiprazole treatment
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Doses were flexibly titrated to between 10 and 30 mg once daily based on the individual needs of the patient as determined by the investigator.
  Other Names: Aripiprazole Orally Disintegrating Tablets; Bosiqing®

SUMMARY:
This study attempts to observe the effectiveness and safety of aripiprazole in hospitalized patients with acute schizophrenia episode, and to compare the different drug regimens that may be involved in order to clarify the characteristics of the population for taking aripiprazole and provide reference for clinical rational drug use.

DETAILED DESCRIPTION:
The control of acute schizophrenia effectively and rapidly will build up the confidence of patients on treatments. These early effects may influence the long-term compliance and prognosis of patients. Aripiprazole is an important drug in first line treatment of schizophrenia. However, at present in China, the application of aripiprazole in some patients with acute schizophrenia is not appropriate, leading to poor control of the positive symptoms of the acute phase.

The purpose of this single-arm, open-label trial is to study the situation of the use of aripiprazole in hospitalized patients with acute schizophrenia episode, and to compare the different drug regimens that may be involved in order to supply important information for optimizing treatment strategies of hospitalized patients characterized by positive symptom.

The hospitalized patients characterized by positive symptom with acute schizophrenia episode were recruited. At the time of enrollment, the demographic, symptomatic and laboratory data was collected. After the completion of the baseline assessment and examination, the patients were given aripiprazole. Clinical evaluation was performed at 1、2、4 and 8 weeks after treatment, including the therapeutic efficacy and adverse drug reactions ,and monitoring of laboratory data.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting International Classification of Diseases (tenth version, ICD-10) criteria for schizophrenia.
* acute episode; inpatients
* Age from 18-65 years old (inclusion), male or female
* PANSS total score at least 70
* scoring ≥ 4 on at least two of the following PANSS items: P1 (delusions), P2 (conceptual disorganisation), P3 (hallucinations), P6 (suspiciousness/persecution) ; and PANSS positive score is higher than PANSS negative score
* Written informed consent

Exclusion Criteria:

* other serious diseases;
* Pregnant or breast feeding women or planning a pregnancy
* Patients in a state of drug-induced malignant syndrome or serious extrapyramidal side effect, or with a history of malignant syndrome or serious extrapyramidal side effect;
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Allergy to Aripiprazole
* History of alcohol or drug abuse or dependence in the past 1-year before screening
* mental retardation; bipolar disorder; major depressive disorder;
* Currently using one kind of antipsychotic drug at a dose that exceeds the recommended maximum dose for two weeks, but no improvement in core symptoms; or currently using two kinds of antipsychotic drugs, at least one of which reaches or exceeds the recommended maximum dose for two weeks, but no improvement in core symptoms; or currently using three kinds of antipsychotic drugs or more;
* Refractory schizophrenia patients who did not respond to treatments of two different type antipsychotics with adequate dose and course
* Patients with clinically significant abnormalities on electrocardiogram or laboratory tests
* Patients with clinically significant abnormalities on liver function (ALT or AST>2 times of higher limit of normal range)
* Patients who had Electroconvulsive Therapy (ECT) in the past 2 months
* Participation in a clinical trial of another drug within 4 weeks prior to study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
PANSS (positive and negative symptoms scale) total score | baseline,8 weeks
  Change from baseline PANSS (positive and negative symptoms scale) total score at 8 weeks
PANSS positive score | baseline,8 weeks
  Change from baseline PANSS positive score at 8 weeks
CGI-S (clinical general impression-severity) | baseline,8 weeks
  Change from baseline CGI-S (clinical general impression-severity) at 8 weeks

SECONDARY OUTCOMES:
PANSS negative score | baseline,8 weeks
  Change from baseline PANSS negative score at 8 weeks
MSQ (Medication Satisfaction Questionnaire)score | baseline,8 weeks
  MSQ score at each assessment time point

OTHER OUTCOMES:
Fasting blood lipids | baseline,4,8 weeks
  Levels of fasting blood lipids
Fasting blood glucose | baseline, 4,8 weeks
  Levels of fasting blood glucose
Serum prolactin | baseline, 4,8 weeks
  Levels of serum prolactin
BMI (body mass index) | baseline,1,2,4,8 weeks
  weight and height will be combined to report BMI in kg/m^2
Waist circumference | baseline,1,2,4,8 weeks
  measurement of waist circumference in centimeters
Hip circumference | baseline,1,2,4,8 weeks
  measurement of hip circumference in centimeters
Occurrence of adverse reactions | baseline,1,2,4,8 weeks
  Occurrence of adverse reactions will be recorded

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - The Fourth People's Hospital of Hefei, Hefei, Anhui
  - Beijing Anding Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing HuiLongGuan Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - The First Haerbin Psychiatric Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Mental Health Center, Wuhan, Hubei
  - 102 Miltary Hospital of China, Changzhou, Jiangsu
  - Shandong Mental Health Center, Jinan, Shandong
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - The Fourth People's Hospital of Chengdu, Chengdu, Sichuan
  - Hangzhou Seventh People's Hospital, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No